CLINICAL TRIAL: NCT06219512
Title: Evaluation of the Clinical Effect of the Formulation of Individualized Exercise Prescription for Hypertension With 6-minute Walking Test (6MWT)
Brief Title: Clinical Effect of Individualized Exercise Prescription for Hypertension With 6-minute Walking Test (6MWT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yang Xi, Doctor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDL2022-23
Record Dates: First submitted 2023-02-22; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: hypertension; Exercise prescription; Intelligent information management; 6-min walking test (6MWT); Cardiopulmonary exercise test (CPET)
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPET exercise prescription group (Experimental): Formulate exercise prescription of cardiopulmonary exercise test (CPET) according to the principle of FITT [frequency, intensity, time and type]
  Interventions: Behavioral: CPET exercise prescription
- 6MWT exercise prescription group (Experimental): Exercise prescription is set according to the recommendation of the Chinese expert consensus on the application of clinical norms of six-minute walking test
  Interventions: Behavioral: 6MWT exercise prescription
- Regular exercise group (Active Comparator): Carry out regular exercise as usual
  Interventions: Behavioral: Regular exercise

INTERVENTIONS:
Behavioral: CPET exercise prescription — Exercise mode: walk Frequency: 5 times/week
  Arms: CPET exercise prescription group
Behavioral: 6MWT exercise prescription — Exercise mode: walk Frequency: 5 times/week
  Arms: 6MWT exercise prescription group
Behavioral: Regular exercise — Regular exercise
  Arms: Regular exercise group

SUMMARY:
Obesity and lack of exercise are one of the reasons for high blood pressure. Exercise can reduce the risk of cardiovascular events by reducing weight and blood pressure. The precise formulation of exercise prescription by cardiopulmonary exercise test (CPET) can effectively control hypertension. Our research group has formulated 50 "exercise prescriptions for hypertension population" in the early stage, but how to further effectively implement them needs to be discussed.

Based on the previous experience of undertaking the project "Exercise Prescription for Hypertensive People" of General Administration of Sport of the People's Republic of China, this research group discussed the important role of intelligent information management in the clinical effect evaluation and effective implementation of exercise prescription for hypertension; To explore the feasibility of making exercise prescription for hypertension based on 6-min walking test, and whether it is not inferior to or equivalent to the accuracy and effectiveness of making exercise prescription by CPET. The relevant results will lay a foundation for exploring the broader adaptation of hypertension exercise prescription to the population.

DETAILED DESCRIPTION:
The 6-minute walking test (6MWT) has good universality and accessibility, and can be used as the basis for formulating exercise prescriptions. According to the consensus of Chinese experts on the application of clinical norms of the six-minute walking test, it is recommended to formulate individualized exercise prescriptions based on the average walking speed of 6MWT calculated from the six-minute walking distance (6MWD), but there is no relevant content about hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obesity; Normal or normal high blood pressure after drug use; Grade 1 hypertension (whether taking medicine or not); Having sports habits; Sports risk is low and medium

Exclusion Criteria:

* ≥ grade 2 Hypertension; High-risk hypertensive patients; Malignant hypertension, secondary hypertension, etc; Serious arrhythmia, heart failure, acute myocardial infarction; Severe stroke, liver and kidney insufficiency; Physical dysfunction and failure to cooperate for various reasons; Unable to conduct CPET; The Types and doses of antihypertensive drugs is still in the process of adjustment

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure, SBP | through study completion, an average of 1 year
  systolic blood pressure (mmHg)
Diastolic blood pressure, DBP | through study completion, an average of 1 year
  diastolic blood pressure (mmHg)
Heart rate, HR | through study completion, an average of 1 year
  Heart rate (beats/min)
Pulse wave velocity, PWV | through study completion, an average of 1 year
  pulse wave velocity
PWV | through study completion, an average of 1 year
  pulse wave velocity
weight | through study completion, an average of 1 year
  weight (kg)
Body mass index, BMI | through study completion, an average of 1 year
  body mass index （kg/m^2）

SECONDARY OUTCOMES:
Blood lipids | through study completion, an average of 1 year
  Triglyceride, total cholesterol, low-density lipoprotein cholesterol
exercise hypertension | through study completion, an average of 1 year
  yes/no
circadian rhythm of blood pressure | through study completion, an average of 1 year
  Ambulatory blood pressure monitoring
anxiety | through study completion, an average of 1 year
  Anxiety score using Generalized Anxiety Disorder (GAD-7). High GAD-7 scores significantly predicted worse state of anxiety: no anxiety,0-4 scores; mild anxiety,5-9 scores; moderate anxiety,10-14 scores; severe anxiety,15-21 scores.
depression | through study completion, an average of 1 year
  Depression score using Patient Health Questionnaire-9 (PHQ-9). High PHQ-9 scores significantly predicted worse state of depression: no depression,0-4 scores; mild depression,5-9 scores; moderate depression,10-14 scores; severe depression,15-27 scores.
use of antihypertensive drugs | through study completion, an average of 1 year
  Record dosage and numbers of antihypertensive drugs using questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xi, Doctor, Study Director — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of patients in the maximum extent

REFERENCES:
- [Background] Pelliccia A, Sharma S, Gati S, Back M, Borjesson M, Caselli S, Collet JP, Corrado D, Drezner JA, Halle M, Hansen D, Heidbuchel H, Myers J, Niebauer J, Papadakis M, Piepoli MF, Prescott E, Roos-Hesselink JW, Graham Stuart A, Taylor RS, Thompson PD, Tiberi M, Vanhees L, Wilhelm M; ESC Scientific Document Group. 2020 ESC Guidelines on sports cardiology and exercise in patients with cardiovascular disease. Eur Heart J. 2021 Jan 1;42(1):17-96. doi: 10.1093/eurheartj/ehaa605. No abstract available. PMID 32860412